CLINICAL TRIAL: NCT00067158
Title: Smoking Cessation Treatment With Transdermal Nicotine Replacement Therapy
Brief Title: Smoking Cessation Treatment With Transdermal Nicotine Replacement Therapy - 1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: New York University (Other)
Responsible Party: Malcome Reid, Ph.D., New York University
Organization: National Institute on Drug Abuse (NIDA) (NIH)
Purpose: Treatment
Other Study IDs: NIDA-CTN-0009-1
Record Dates: First submitted 2003-08-12; First posted 2003-08-13 (Estimated); Last update posted 2017-01-12 (Estimated); Status verified 2010-04

CONDITIONS: Tobacco Use Disorder
Keywords: nicotine dependence
MeSH Terms: conditions — Tobacco Use Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: nicotine transdermal system

SUMMARY:
The purpose of this study is to look at how feasible it is to incorporate a state-of-the-art smoking cessation treatment program into community substance abuse treatment programs and its impact on substance abuse and cigarette smoking.

ELIGIBILITY:
Inclusion Criteria:

* Patient is alcohol or drug dependent, in Outpatient Drug-Free or Opiate Substitute program and is interested in quitting smoking

Exclusion Criteria:

* Patient is psychotic
* Use of smokeless tobacco
* Use of other smoking cessasation product
* Pregnancy
* Patient has hyper-tension, heart problems, or skin condition

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 585
Dates: Start 2003-04; Primary Completion 2004-07 (Actual); Study Completion 2004-07 (Actual)

PRIMARY OUTCOMES:
Drug use
Smoking Cessation

CONTACTS AND LOCATIONS:
Overall Officials: Malcolm Reid, Ph.D., Principal Investigator — New York University
Locations (13):
- United States (13):
  - Matrix Institute on Addictions, Los Angeles, California
  - Tarzana Treatment Center, Tarzana, California
  - SPECTRUM, Miami, Florida
  - Center for Drug Free Living, Orlando, Florida
  - Chelsea Arbor Addictions Treatment Center, Ann Arbor, Michigan
  - Psychiatry and Behavioral Medicine Professionals I, Detroit, Michigan
  - Narco Freedom (Bridge Plaza), Long Island City, New York
  - St. Luke's Roosevelt Hospital Center, New York, New York
  - St. Luke's Roosevelt Hospital Center, Womens, New York, New York
  - Mount Sinai Medical Center, New York, New York
  - Piedmont Behavioral Healthcare, Concord, North Carolina
  - Coastal Horizons Center, Inc., Wilmington, North Carolina
  - Behavioral Health Services of Pickens County, Pickens, South Carolina

REFERENCES:
- See also: Data Elements — http://www.ctndatashare.org/protocol-ctndatashare/new-protocols/nida-ctn-0009